CLINICAL TRIAL: NCT07293832
Title: The Impact of Sympathetic Drive Control With Cardio-Selective Beta-Blockers on Infarct Size After Acute Myocardial Infarction
Brief Title: Impact of Cardio-Selective Beta-Blockers on Infarct Size After Acute Myocardial Infarction
Acronym: BLOCK-AMI
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Nikolaos Fragakis, Professor of Cardiology, Aristotle University Of Thessaloniki
Other Study IDs: 22/28-3-2023_5123
Record Dates: First submitted 2025-11-25; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: STEMI
Keywords: beta-blocker
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intravenous BB (receiving landiolol) or p.o. BB: STEMI patients receiving beta-blocker

SUMMARY:
Introduction: The effect of intravenous beta-blockers on the extent of the necrotic area, after primary percutaneous transluminal coronary angioplasty (PTCA), for acute myocardial infarction is not well established.

Purpose: The present study aims to investigate, whether the early intravenous administration of landiolol, a highly cardioselective b-blocker, reduces the extent of the necrotic area after ST-elevation myocardial infarction (STEMI).

Methods: This prospective observational cohort study will enroll patients presenting with STEMI, who undergo primary PCI and receive either intravenous landiolol or standard oral β-blocker therapy, in accordance with current European Society of Cardiology (ESC) guidelines. Eligibility will be determined by predefined inclusion and exclusion criteria. Treatment selection will be based solely on the clinical judgment of the attending cardiologist, without randomization.

Results: Final infarct size will be quantified by cardiac magnetic resonance imaging (CMR) performed at least three months after the STEMI to minimize edema-related overestimation. Myocardial function will be assessed during hospitalization using transthoracic echocardiography, including measurement of global longitudinal strain (GLS). Additional data will include serial high-sensitivity troponin and creatine phosphokinase (CPK) measurements, 24-hour continuous electrocardiographic monitoring for arrhythmia burden, and predefined safety outcomes collected throughout hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients with electrocardiogram showing ST-segment elevation ≥2 mm in 2 or more contiguous leads for more than 30 minutes
* Estimated time from symptom onset to reperfusion ≤12 hours
* Patients scheduled to undergo primary angioplasty
* Patients who have signed a consent form

Exclusion Criteria:

* Patients receiving chronic medication with beta-adrenergic blockers
* Patients with a previous myocardial infarction
* Persistent systolic blood pressure <90 mmHg
* Persistent heart rate <55 beats per minute
* Patients with Killip class III (acute pulmonary edema) or IV (cardiogenic shock) on initial examination
* 12-lead electrocardiogram with PR interval >200 milliseconds
* 12-lead electrocardiogram showing second- or third-degree atrioventricular block
* Bronchospasm requiring bronchodilator treatment
* Possible pregnancy or postpartum period
* Inability or refusal to sign the consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with STEMI presenting to Hippokration General Hospital of Thessaloniki will be evaluated for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Infarct Size (CMR) | CMR will be done at least 3months after the myocardial infarction.
  This measurement represents one of the two co-primary outcomes of the study. Infarct size will be quantified by cardiac magnetic resonance imaging (CMR) and expressed in grams. CMR will be performed at least 3 months after the myocardial infarction to minimize the influence of myocardial edema.
Global Longitudinal Strain (GLS) | Within the first 5 days after acute myocardial infarction.
  This measurement represents one of the two co-primary outcomes of the study. Left ventricular global longitudinal strain will be assessed by transthoracic echocardiography during hospitalization to evaluate myocardial systolic function.

SECONDARY OUTCOMES:
Arrhythmia burden | First 24 hours after percutaneous coronary intervention
  Arrhythmia burden will be quantified from continuous telemetry monitoring during the first 24 hours after PCI. The arrhythmia burden will be expressed as a composite index integrating the following components obtained from the same monitoring period:
  * frequency of non-sustained ventricular tachycardia (NSVT) episodes (≥3 consecutive ventricular beats lasting <30 seconds),
  * frequency of ventricular tachycardia (VT) episodes (≥3 consecutive ventricular beats lasting ≥30 seconds),
  * cumulative duration (in seconds) of all NSVT/VT episodes, and
  * total number of ventricular ectopic beats recorded during NSVT/VT events. All components will be analyzed collectively as quantitative descriptors of the overall arrhythmia burden.
Biomarkers of myocardial injury - Peak hs-Troponin I (ng/mL) | At the diagnosis of STEMI, and subsequently at 1 hour, 24 hours, 48 hours, and 72 hours.
  Serial measurements of hs-troponin concentrations will be performed. Hs-troponin will be measured in ng/ml. Reported summary measure will include the peak value from the scheduled samples. Samples are obtained as part of routine clinical care and analyzed by the site laboratory.
Safety Outcome - Number of participants with Cardiogenic shock | From admission until hospital discharge (up to 10 days).
  Number of participants who develop cardiogenic shock during hospitalization, defined as sustained hypotension accompanied by clinical or laboratory evidence of end-organ hypoperfusion and requiring initiation of inotropic support.
Safety Outcome - Number of participants with Symptomatic bradycardia / conduction abnormalities | From admission until hospital discharge (up to 10 days).
  Number of participants with new or worsened symptomatic bradycardia (heart rate <55 bpm with symptoms) or new conduction disturbances (e.g., new second- or third-degree AV block), documented by ECG or telemetry.
Safety Outcome - Number of participants with Hypotension | From admission until hospital discharge (up to 10 days).
  Number of participants who develop hypotension defined as systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg, as recorded in observations.
Safety Outcome - Number of participants with recurrence of myocardial infarction or angina | From admission until hospital discharge (up to 10 days).
  Number of participants with documented recurrent myocardial infarction or recurrent ischemic chest pain (angina) requiring medical evaluation or intervention.
Safety Outcome - Number of participants with new or worsened Heart Failure | From admission until hospital discharge (up to 10 days).
  Number of participants who develop sudden worsening of chronic heart failure (HF) or new-onset HF with congestion requiring therapy or prolongation of hospital stay.
Safety Outcome - Number of participants with cardiovascular death (In-Hospital Cardiovascular Mortality) | From admission until hospital discharge (up to 10 days).
  Number of participants with cardiovascular death occurring during the hospitalization, defined as death resulting from acute myocardial infarction, arrhythmia, cardiogenic shock, progressive heart failure, sudden cardiac death, death due to cardiovascular procedures (e.g., PCI complications), or death from other confirmed cardiovascular pathology such as aortic dissection, acute valvular failure, or pulmonary embolism.
Biomarkers of myocardial injury - Area under the curve for Creatine phosphokinase (ng·h/mL) | Baseline to 72 hours.
  Area under the curve for creatinine phosphokinase (CPK) calculated using the trapezoidal rule from serial CPK measurements.
Biomarkers of myocardial injury - Area Under the Curve for hs-Troponin I (ng·h/mL) | Baseline to 72 hours.
  Area under the curve calculated using the trapezoidal rule from serial hs-Troponin I measurements. Samples are obtained as part of routine clinical care and analyzed by the site laboratory.
Biomarkers of myocardial injury - Peak creatinine phosphokinase (U/L) | At the diagnosis of STEMI, and subsequently at 1 hour, 24 hours, 48 hours, and 72 hours.
  Serial measurements of creatinine phosphokinase (CPK) concentrations will be performed. CPK will be measured in U/L. Reported summary measure will include the peak value from the scheduled samples. Samples are obtained as part of routine clinical care and analyzed by the site laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Fragakis, Professor fo Cardiology, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Hippokration General Hospital of Thessaloniki, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nasoufidou A, Bantidos MG, Stachteas P, Moysidis DV, Mitsis A, Fyntanidou B, Kouskouras K, Karagiannidis E, Karamitsos T, Kassimis G, Fragakis N. The Role of Landiolol in Coronary Artery Disease: Insights into Acute Coronary Syndromes, Stable Coronary Artery Disease and Computed Tomography Coronary Angiography. J Clin Med. 2025 Jul 23;14(15):5216. doi: 10.3390/jcm14155216. PMID 40806838